CLINICAL TRIAL: NCT03742050
Title: A Placebo-controlled Trial of Percutaneous Coronary Intervention for the Relief of Stable Angina
Acronym: ORBITA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Basildon and Thurrock Hospitals NHS FoundationTrust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18SM4531
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Stable Angina
Keywords: Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Percutaneous Coronary Intervention; Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous coronary intervention (Active Comparator): Percutaneous coronary intervention with drug-eluting stents and modern techniques
  Interventions: Procedure: Percutaneous coronary intervention
- Placebo percutaneous coronary intervention (Placebo Comparator): Placebo percutaneous coronary intervention
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention with drug-eluting stents aiming to achieve complete revascularisation
  Other Names: Coronary angioplasty

SUMMARY:
ORBITA-2 is a double blinded randomised placebo-controlled trial comparing the effects of coronary angioplasty versus placebo procedure on symptoms of stable angina without background anti-anginal therapy. Follow-up will be at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

ORBITA-2 will enrol patients who meet all 3 of the following criteria:

1. Angina or angina-equivalent symptoms
2. Anatomical evidence of significant coronary stenosis in at least one vessel, either: a. Invasive diagnostic coronary angiogram indicating ≥ 70% stenosis b. CT coronary angiography indicating ≥ 90% stenosis
3. Evidence of ischaemia, arising from at least one of the following options:

   1. Positive dobutamine stress echocardiography
   2. Positive cardiac MRI perfusion scan
   3. Positive nuclear medicine myocardial perfusion scan
   4. Invasive pressure wire assessment suggestive of ischaemia, as judged by the interventional cardiologist, at the time of diagnostic angiogram or research angiogram

Exclusion Criteria:

1. Age younger than 18
2. Age older than 85
3. Recent acute coronary event
4. Previous coronary artery bypass graft surgery
5. Significant left main stem coronary disease
6. Chronic total occlusion in the target vessel
7. Contraindication to percutaneous coronary intervention or drug-eluting stent implantation
8. Contraindication to antiplatelet therapy
9. Severe valvular disease
10. Severe LV systolic impairment
11. Severe respiratory disease
12. Life expectancy less than 2 years, pregnancy, unable to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Change in angina symptom score between groups | 12 weeks

SECONDARY OUTCOMES:
Change in treadmill exercise time | 12 weeks
Angina severity as assessed by Canadian Cardiovascular Society class | 12 weeks
Physical limitation, angina stability, quality of life, angina frequency, freedom from angina as assessed with the Seattle Angina Questionnaire | 12 weeks
Quality of life as assessed with the EQ-5D-5L questionnaire | 12 weeks
Change in dobutamine stress echocardiography score | 12 weeks
Need for anti-anginal medication introduction and up-titration | 12 weeks
Admission for acute coronary syndrome or unscheduled coronary angiography | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darrel Francis, MRCP, Study Chair — Imperial College London; Christopher A Rajkumar, Study Director — Imperial College London; Rasha Al-Lamee, Principal Investigator — Imperial College London
Locations (8):
- United Kingdom (8):
  - Basildon and Thurrock Hospitals NHS Foundation Trust, Basildon
  - Royal Bournemouth Hospital, Bournemouth
  - Wycombe Hospital, High Wycombe
  - Imperial College Healthcare NHS Trust, London
  - Royal Free Hospital, London
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire NHS Foundation Trust, Reading
  - Harefield Hospital, Uxbridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simader FA, Rajkumar CA, Foley MJ, Ahmed-Jushuf F, Chotai S, Chiew K, Naderi Z, Davies JR, Keeble TR, O'Kane PD, Haworth P, Nijjer SS, Howard JP, Cole G, Harrell FE Jr, Francis DP, Shun-Shin MJ, Al-Lamee RK; ORBITA-2 Investigators. Association Between Age and PCI Effectiveness in Stable CAD: Secondary Analysis of ORBITA-2. J Am Coll Cardiol. 2026 Jan 27;87(3):253-265. doi: 10.1016/j.jacc.2025.10.086. PMID 41603507
- [Derived] Foley MJ, Rajkumar CA, Ahmed-Jushuf F, Simader F, Chotai S, Seligman H, Macierzanka K, Davies JR, Keeble TR, O'Kane P, Haworth P, Routledge H, Kotecha T, Clesham G, Williams R, Din J, Nijjer SS, Curzen N, Sinha M, Petraco R, Spratt J, Sen S, Cole GD, Harrell FE Jr, Howard JP, Francis DP, Shun-Shin MJ, Al-Lamee R; ORBITA-2 Investigators. Fractional Flow Reserve and Instantaneous Wave-Free Ratio as Predictors of the Placebo-Controlled Response to Percutaneous Coronary Intervention in Stable Coronary Artery Disease. Circulation. 2025 Jan 21;151(3):202-214. doi: 10.1161/CIRCULATIONAHA.124.072281. Epub 2024 Oct 27. PMID 39462291
- [Derived] Rajkumar CA, Foley MJ, Ahmed-Jushuf F, Nowbar AN, Simader FA, Davies JR, O'Kane PD, Haworth P, Routledge H, Kotecha T, Gamma R, Clesham G, Williams R, Din J, Nijjer SS, Curzen N, Ruparelia N, Sinha M, Dungu JN, Ganesananthan S, Khamis R, Mughal L, Kinnaird T, Petraco R, Spratt JC, Sen S, Sehmi J, Collier DJ, Sohaib A, Keeble TR, Cole GD, Howard JP, Francis DP, Shun-Shin MJ, Al-Lamee RK; ORBITA-2 Investigators. A Placebo-Controlled Trial of Percutaneous Coronary Intervention for Stable Angina. N Engl J Med. 2023 Dec 21;389(25):2319-2330. doi: 10.1056/NEJMoa2310610. Epub 2023 Nov 11. PMID 38015442
- [Derived] Nowbar AN, Rajkumar C, Foley M, Ahmed-Jushuf F, Howard JP, Seligman H, Petraco R, Sen S, Nijjer SS, Shun-Shin MJ, Keeble TR, Sohaib A, Collier D, McVeigh P, Harrell FE, Francis DP, Al-Lamee RK. A double-blind randomised placebo-controlled trial of percutaneous coronary intervention for the relief of stable angina without antianginal medications: design and rationale of the ORBITA-2 trial. EuroIntervention. 2022 Apr 22;17(18):1490-1497. doi: 10.4244/EIJ-D-21-00649. PMID 35156616